CLINICAL TRIAL: NCT02412111
Title: A Phase 3, Randomized, Double-Blind, Ivacaftor-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of VX-661 in Combination With Ivacaftor in Subjects Aged 12 Years and Older With Cystic Fibrosis, Heterozygous for the F508del-CFTR Mutation and a Second CFTR Allele With a Gating Defect That Is Clinically Demonstrated to be Ivacaftor Responsive
Brief Title: A Phase 3 Study of Tezacaftor (VX-661) in Combination With Ivacaftor (VX-770) in Subjects Aged 12 Years and Older With Cystic Fibrosis (CF), Who Have One F508del-CFTR Mutation and a Second Mutation That Has Been Demonstrated to be Clinically Responsive to Ivacaftor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX14-661-109
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor; tezacaftor, ivacaftor drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ivacaftor (Run-in Period) (Experimental): Ivacaftor 150 milligram (mg) tablet orally every 12 hours for 4 weeks.
  Interventions: Drug: Ivacaftor
- VX-661 + Ivacaftor (Active comparator period) (Experimental): VX-661 100 mg and ivacaftor 150 mg fixed-dose combination tablet orally once daily in the morning and ivacaftor 150 mg tablet orally once daily in the evening for 8 weeks.
  Interventions: Drug: Ivacaftor; Drug: Tezacaftor/Ivacaftor
- Ivacaftor monotherapy (Active comparator period) (Active Comparator): Ivacaftor 150 mg tablet orally every 12 hours as monotherapy for 8 weeks.
  Interventions: Drug: Ivacaftor

INTERVENTIONS:
Drug: Ivacaftor
  Other Names: VX-770
Drug: Tezacaftor/Ivacaftor
  Other Names: VX-661/VX-770
  Arms: VX-661 + Ivacaftor (Active comparator period)

SUMMARY:
This is a Phase 3, randomized, double-blind, ivacaftor-controlled, parallel-group, multicenter study of tezacaftor in combination with ivacaftor in subjects aged 12 years and older with CF who are heterozygous for the F508del-CFTR mutation and a second CFTR allele with a gating defect that is clinically demonstrated to be ivacaftor responsive.

ELIGIBILITY:
Inclusion Criteria:

* Heterozygous for F508del-CFTR mutation and a second CFTR allele with a gating defect that is clinically demonstrated to be ivacaftor responsive
* FEV1 ≥40% and ≤90% of predicted normal for age, sex, and height during screening
* Stable CF disease as judged by the investigator.

Exclusion Criteria:

* History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Pregnant and nursing females (females of childbearing potential must have a negative pregnancy test at Screening and Week -4 Visits).
* Sexually active subjects of reproductive potential who are not willing to follow the contraception requirements

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (68):
- United States (33):
  - Birmingham, Alabama
  - Oakland, California
  - San Diego, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Augusta, Georgia
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Manchester, New Hampshire
  - Morristown, New Jersey
  - New Brunswick, New Jersey
  - Albany, New York
  - New York, New York
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - Morgantown, West Virginia
- Australia (5):
  - Chermside
  - Clayton
  - Melbourne
  - South Brisbane
  - Westmead
- Innsbruck, Austria
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Canada (3):
  - Calgary
  - Toronto
  - Vancouver
- Paris, France
- Germany (8):
  - Dresden
  - Erlangen
  - Essen
  - Frankfurt
  - Giessen
  - Heidelberg
  - Jena
  - München
- Ireland (2):
  - Cork
  - Dublin
- Italy (3):
  - Bari
  - Milan
  - Roma
- United Kingdom (9):
  - Belfast
  - Birmingham
  - Cardiff
  - Glasgow
  - Leeds
  - London
  - Manchester
  - Newcastle
  - Southampton

REFERENCES:
- [Derived] McKone EF, DiMango EA, Sutharsan S, Barto TL, Campbell D, Ahluwalia N, Higgins M, Owen CA, Tullis E. A phase 3, randomized, double-blind, parallel-group study to evaluate tezacaftor/ivacaftor in people with cystic fibrosis heterozygous for F508del-CFTR and a gating mutation. J Cyst Fibros. 2021 Mar;20(2):234-242. doi: 10.1016/j.jcf.2020.11.003. Epub 2020 Dec 16. PMID 33339768

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 periods: an Ivacaftor Run-in Period and an Active Comparator Treatment Period. Participants were randomized in a ratio of 1:1 to receive either VX-661/ivacaftor combination therapy or ivacaftor monotherapy for 8 weeks during the Active Comparator Treatment Period after completion of 4 weeks Ivacaftor Run-in Period.
Period: Ivacaftor Run-in Period (4 Weeks)
Arm/Group | Ivacaftor (Run-in Period) | VX-661 + Ivacaftor (Active Comparator Period) | Ivacaftor Monotherapy (Active Comparator Period)
Started | 156 | 0 | 0
Completed | 153 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Did not meet eligibility criteria | 1 | 0 | 0
Not completed — Participants refused further dosing | 2 | 0 | 0
Period: Active Comparator Period (8 Weeks)
Arm/Group | Ivacaftor (Run-in Period) | VX-661 + Ivacaftor (Active Comparator Period) | Ivacaftor Monotherapy (Active Comparator Period)
Started (Two participants who completed the Run-in period did not enter the active comparator period.) | 0 | 76 | 75
Full Analysis Set | 0 | 76 | 74
Completed | 0 | 75 | 69
Not Completed | 0 | 1 | 6
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Participants refused further dosing | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other non-compliance | 0 | 1 | 0
Not completed — Other | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who were included in Full Analysis Set for active comparator period (all randomized participants who have received at least 1 dose of blinded study drug during the active comparator treatment period.)
Groups:
- Total: Total of all reporting groups
Arm/Group | VX-661 + Ivacaftor (Active Comparator Period) | Ivacaftor Monotherapy (Active Comparator Period) | Total
Number analyzed (Participants) | 76 | 74 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (13.1) | 31.8 (11.1) | 32.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 34 | 66
  Male | 44 | 40 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 76 | 72 | 148
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 73 | 72 | 145
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Through Week 8
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Through Week 8
Population: Full Analysis Set was defined as all randomized participants who have received at least 1 dose of blinded study drug during the active comparator treatment period. Here "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percent predicted of FEV1
Arm/Group | VX-661 + Ivacaftor (Active Comparator Period) | Ivacaftor Monotherapy (Active Comparator Period)
Number analyzed (Participants) | 76 | 72
Percent predicted of FEV1 | 0.5 (0.4) | 0.2 (0.4)
Statistical Analysis 1: Comparison: VX-661 + Ivacaftor (Active Comparator Period) vs Ivacaftor Monotherapy (Active Comparator Period); Test type: Superiority; p = 0.5846, Mixed Model for Repeated Measures (MMRM); Least Square (LS) mean difference = 0.3, 95% CI 2-sided [-0.8 to 1.4]

2. Secondary Outcome: Relative Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Through Week 8
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Through Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | VX-661 + Ivacaftor (Active Comparator Period) | Ivacaftor Monotherapy (Active Comparator Period)
Number analyzed (Participants) | 76 | 72
Percent change | 1.3 (0.6) | 0.5 (0.6)
Statistical Analysis 1: Comparison: VX-661 + Ivacaftor (Active Comparator Period) vs Ivacaftor Monotherapy (Active Comparator Period); Test type: Superiority; p = 0.3860, Mixed models Repeated Measures (MMRM); Least square mean difference = 0.8, 95% CI 2-sided [-1.0 to 2.6]

3. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score From Baseline Through Week 8
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: Baseline, Through Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | VX-661 + Ivacaftor (Active Comparator Period) | Ivacaftor Monotherapy (Active Comparator Period)
Number analyzed (Participants) | 76 | 73
units on a scale | 0.7 (1.3) | -2.1 (1.3)
Statistical Analysis 1: Comparison: VX-661 + Ivacaftor (Active Comparator Period) vs Ivacaftor Monotherapy (Active Comparator Period); Test type: Superiority; p = 0.1236, Mixed models Repeated Measures (MMRM); Least square mean difference = 2.8, 95% CI 2-sided [-0.8 to 6.4]

4. Secondary Outcome: Absolute Change From Baseline in Sweat Chloride Through Week 8
Description: Sweat samples were collected using an approved collection device.
Time Frame: Baseline, Through Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter
Arm/Group | VX-661 + Ivacaftor (Active Comparator Period) | Ivacaftor Monotherapy (Active Comparator Period)
Number analyzed (Participants) | 74 | 70
Millimoles per liter | -7.9 (1.7) | -2.1 (1.8)
Statistical Analysis 1: Comparison: VX-661 + Ivacaftor (Active Comparator Period) vs Ivacaftor Monotherapy (Active Comparator Period); Test type: Superiority; p = 0.0216, Mixed models Repeated Measures (MMRM); Least square mean difference = -5.8, 95% CI 2-sided [-10.7 to -0.9]

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to Week 16
Population: The Safety Set included all participants who received at least 1 dose of study drug during Ivacaftor (Run-in period) and active comparator treatment period.
Measure: Number; unit: Participants
Arm/Group | Ivacaftor (Run-in Period) | VX-661 + Ivacaftor (Active Comparator Period) | Ivacaftor Monotherapy (Active Comparator Period)
Number analyzed (Participants) | 156 | 76 | 75
Participants
  Participants with AEs | 66 | 50 | 54
  Participants with SAEs | 2 | 4 | 7

6. Secondary Outcome: Trough Plasma Concentrations (Ctrough) of VX-661, VX-661 Metabolites (M1-VX-661), Ivacaftor (IVA) and IVA Metabolite (M1-IVA)
Time Frame: Predose on Week -2 for Run-in period; Pre-dose on Week 2 for Active comparator period
Population: Pharmacokinetic (PK) set included participants who received study drug and had PK assessment. Here 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome. "Number Analyzed=0" indicates no participants were analyzed for specified categories because VX-661 was not administered in the specified arms.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Ivacaftor (Run-in Period) | VX-661 + Ivacaftor (Active Comparator Period) | Ivacaftor Monotherapy (Active Comparator Period)
Number analyzed (Participants) | 143 | 75 | 68
nanogram per milliliter (ng/mL)
  IVA | 812 (615) | 1000 (742) | 740 (464)
  M1-IVA | 1590 (956) | 1830 (1010) | 1450 (828)
  VX-661: number analyzed (Participants) | 0 | 75 | 0
  VX-661 |  | 2520 (1490) |
  M1-VX-661: number analyzed (Participants) | 0 | 75 | 0
  M1-VX-661 |  | 4870 (1750) |

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Arm/Group | Ivacaftor (Run-in Period) | VX-661 + Ivacaftor (Active Comparator Period) | Ivacaftor Monotherapy (Active Comparator Period)
All-Cause Mortality (participants affected / at risk) | 0/156 | 0/76 | 0/75
Serious Adverse Events (participants affected / at risk) | 2/156 | 4/76 | 7/75
Other Adverse Events (participants affected / at risk) | 24/156 | 25/76 | 32/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ivacaftor (Run-in Period) (N=156) | VX-661 + Ivacaftor (Active Comparator Period) (N=76) | Ivacaftor Monotherapy (Active Comparator Period) (N=75)
Human rhinovirus test positive (Investigations) | 1 | 0 | 0
Idiopathic intracranial hypertension (Nervous system disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 2 | 5
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ivacaftor (Run-in Period) (N=156) | VX-661 + Ivacaftor (Active Comparator Period) (N=76) | Ivacaftor Monotherapy (Active Comparator Period) (N=75)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 12 | 12
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 4
Dizziness (Nervous system disorders) | 2 | 4 | 0
Fatigue (General disorders) | 4 | 5 | 2
Nausea (Gastrointestinal disorders) | 3 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 6 | 4
Viral upper respiratory tract infection (Infections and infestations) | 1 | 4 | 6
Headache (Nervous system disorders) | 10 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1)first multi-center publication, (2)if sponsor elects not to publish the results, or(3)18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.

DOCUMENTS (2):
  • Study Protocol (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT02412111/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT02412111/SAP_001.pdf